CLINICAL TRIAL: NCT02227004
Title: Safety of Clinically Indicated Magnetic Resonance Imaging in Patients With Permanent Pacemakers (PPM) and Implanted Cardioverter Defibrillators
Brief Title: Safety of Magnetic Resonance Imaging in Patients With Pacemakers and Defibrillators
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00051707
Record Dates: First submitted 2014-08-20; First posted 2014-08-27 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Conditions Requiring Diagnostic Evaluation
Keywords: MRI; Magnetic Resonance Imaging; pacemakers; ICD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Males and females 9 years or older weighing at least 80 lbs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI in patients with Pacemaker or ICD: Perform MRI in patients with pacemaker or ICD and evaluate patient and device safety
  Interventions: Diagnostic Test: Perform MRI in patients with pacemaker or ICD

INTERVENTIONS:
Diagnostic Test: Perform MRI in patients with pacemaker or ICD — Perform MRI in patients with pacemaker or ICD

SUMMARY:
Pacemakers and ICD's have traditionally been accepted as contraindications to MRI due to safety concerns. Recent work in our laboratory as well as our pilot study of approximately 500 patients has shown the safety of most contemporary implanted rhythm management devices in the MRI environment given appropriate precautions. Because the investigators have completed testing in animals weighing as little as 80 lbs. without incident, the investigators feel they can safely image children at this weight or greater (Circulation 2004; 110:475-482).

The goal of this study is to expand on our pilot study and to develop a protocol, consistent with the Department of Health and Human Services (DHHS) requirements, that will increase our safety experience with clinically indicated MR imaging in patients with implanted cardiac pacemakers and ICD's.

This is a cohort study. One thousand seven hundred patients with a clinical need for MRI will be recruited. Risks and Benefits associated with Magnetic Resonance (MR) imaging in the setting of implantable devices will be discussed and informed consent obtained. The type of device and leads will be ascertained. Patients will be monitored by a physician or a Registered Nurse (RN) with ACLS certification and familiarity with ICD/Pacemaker programming during the study. When imaging children who meet age and weight criteria, a physician will be present during the entire study. Fellow and attending radiology and electrophysiology support will be available in house in all cases.

Standard device testing including battery voltages, thresholds, sensing and lead impedances will be measured.

DETAILED DESCRIPTION:
The primary objective of this study is to develop a protocol, consistent with DHHS/ Center for Medicare and Medicaid Services (CMS) guidelines and requirements to further document safety in clinically indicated MR imaging in patients with implanted cardioverter defibrillators (ICD's) and pacemakers.

MRI's will be conducted on patients who require a clinically indicated MRI only. All studies will be done in the 1.5 Tesla MRI unit. ECG monitoring pads will be placed on the patients for the duration of the study. An external defibrillator and Advance Cardiovascular Life Support (ACLS) drugs will be on hand. Heart rate, blood pressure, O2 saturation will also be monitored non-invasively throughout the study. All devices will undergo a complete interrogation prior to imaging. Parameters such as atrial and ventricular pacing thresholds, R and P wave amplitudes, lead impedance, and battery status will be measured and recorded. PPMs will be programmed to an asynchronous mode if dependent and to an inhibited mode in patients without pacemaker dependence.

The pacemaker function of ICD's in pacemaker independent patients will be programmed to ventricular inhibited (VVI) mode at 50 bpm. Pacemaker dependant patients with ICDs will be excluded.

In addition, there is a theoretical concern that patients who have capped or abandoned leads in their chest may be at risk for heating. While there is little or no objective data to support this concern, given this theoretical concern, patients in this category will only be admitted to the study if the referring physician deems the MRI critical and after the PI has carefully considered the risk/benefit ration for each patient who falls in to this category.

Similarly, there historically has also been a concern that newly implanted leads (<4 weeks) are at risk for lead to dislodgement d/t possible torque from the MRI environment. This too is only a theoretical concern and there is little or no scientific evidence to support this claim. Nevertheless, patients with newly implanted pacemaker/ICD leads will be considered by the PI for protocol inclusion only if the referring physician deems the MRI to be critical and after considering the risk/benefit to each individual patient.

After the appropriate MRI protocol for each MRI patient's unique condition has been completed, the device will be re-programmed to its original settings and completely interrogated to detect any changes in device performance.

ELIGIBILITY:
Inclusion Criteria:

Patients with an absolute clinical need for MR imaging and PPM (year 1996 model or later) or ICD's (year 2000 or later)

-

Exclusion Criteria:

Inclusion: Patients with an absolute clinical need for MR imaging and PPM (year 1996 model or later) or ICD's (year 2000 or later)

Exclusion:

* Patients with pacemaker models before 1996 and ICD models before year 2000.
* Pacemaker defendant patients with ICD.
* Patients who weighing less than 80 lbs.
* Patients less than 9 years old
* Patients who complete the MRI standard screening form and are deemed inappropriate for MRI for any reason
* Pregnant patients will be excluded in their first trimester and will not get gadolinium at any time during their pregnancy
* Patient with abandoned/capped leads or leads implanted <4 weeks unless the procedure is deemed critical by the referring physician and approved by the PI

Ages: 9 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females 9 years old or greater weighing more than 80 lbs who require a clinically indicated MRI
Sampling Method: Non-Probability Sample
Enrollment: 1275 (Actual)
Dates: Start 2011-12-30 (Actual); Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

PRIMARY OUTCOMES:
Patient safety and device malfunction during or after MRI | post MRI
  Device function will be assessed by comparing pre-vs. post MRI battery voltage, impedance, sensing and capture thresholds

CONTACTS AND LOCATIONS:
Overall Officials: Henry R. Halperin, M.D.,M.A., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Blalcok 5 MRI, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nazarian S, Hansford R, Rahsepar AA, Weltin V, McVeigh D, Gucuk Ipek E, Kwan A, Berger RD, Calkins H, Lardo AC, Kraut MA, Kamel IR, Zimmerman SL, Halperin HR. Safety of Magnetic Resonance Imaging in Patients with Cardiac Devices. N Engl J Med. 2017 Dec 28;377(26):2555-2564. doi: 10.1056/NEJMoa1604267. PMID 29281579
- See also: PubMed Citation #1 — https://pubmed.ncbi.nlm.nih.gov/29281579/